CLINICAL TRIAL: NCT00857857
Title: A Randomised, Placebo-controlled, Incomplete Block, Three-way Cross-over Study to Evaluate the Effect of Treatment With Repeat Inhaled Doses of GW870086X on the Allergen-induced Early and Late Asthmatic Response in Subjects With Mild Asthma
Brief Title: A Study to Evaluate the Effect of GW870086X on Allergen Challenge in Mild Asthmatics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 110762
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Results first posted 2018-02-20 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2017-08

CONDITIONS: Asthma
Keywords: asthma; late phase response; allergen; challenge; GW870086X
MeSH Terms: conditions — Asthma | interventions — GW870086X

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 13 day repeat dose (Experimental)
  Interventions: Drug: GW870086X; Drug: FP; Drug: Placebo

INTERVENTIONS:
Drug: GW870086X — Investigational product
Drug: FP — Positive control
Drug: Placebo — Placebo control

SUMMARY:
The study will measure the early and late asthamtic response using an allergen challenge. This study will evaluate the safety and patients tolerance to repeat inhaled doses of GW870086X using a number of clinical and biological markers.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects between 18 and 65 years of age inclusive.
* Male subjects must agree to use one of the contraception methods listed in Section 8. This criterion must be followed from the time of the first dose of study medication until 90-95 hours post-last dose.
* BMI within the range 19.0 - 29.0 kg/m2 (inclusive).
* Liver function tests (bilirubin, AST, ALT) within normal laboratory parameters at screening.
* Documented history of bronchial asthma, first diagnosed at least 6 months prior to the screening visit and currently being treated only with intermittent short-acting beta -agonist therapy by inhalation.
* Pre-bronchodilator FEV1 >65% of predicted at screening.
* No history of smoking within 6 months of the start of the study, and with a total pack year history of <= 10 pack years
* Demonstration of a positive wheal and flare reaction (>= 3 mm relative to negative control) to at least one allergen from a battery of allergens (including but not limited to house dust mite, grass pollen, cat dander, hazel, horse and birch) on skin prick testing at screening, or within 12 months of study start.
* Screening allergen challenge demonstrates that the subject experiences both an early and late asthmatic response. The early asthmatic response must include a fall in FEV1 of >= 20% from the post saline value, on at least one occasion, between 5 and 30 minutes after the final concentration of allergen. The late asthmatic response must include a fall in FEV1 of >= 15% from the post saline value, on at least three occasions, two of which must be consecutive, between 4 and 10 hours after the final concentration of allergen.
* Reproducible allergen challenge at screening (confirmation of the dose ascending allergen challenge by a bolus allergen challenge at least 14 days later).
* Sensitivity to methacholine with a provocative concentration of methacholine resulting in a 20% fall in FEV1 (PC20 methacholine) of <8 mg/mL at screening.
* Subjects who are able to produce acceptable induced sputum samples (as defined in the Study Procedures Manual).
* Be able to give written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Single QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, bronchiectasis or pulmonary fibrosis).
* Clinically significant abnormalities in safety laboratory analysis at screening.
* Subject has known history of hypertension or is hypertensive at screening. Hypertension at screening is defined as persistent systolic BP >140mmHg or diastolic BP > 90mmHg.
* Respiratory tract infection and/or exacerbation of asthma within 4 weeks prior to the first dose of study medication.
* History of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnoea, respiratory arrest and/or hypoxic seizures.
* Administration of oral, injectable or dermal steroids within 4 weeks or intranasal and/or inhaled steroids within 2 week of the screening visit.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as:

an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males). One unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.

* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety. Paracetamol is an exception and will be permitted at daily doses of up to 4 g from screening to follow-up.
* Has taken Xanthines (including theophylline, but not including caffeine), anticholinergics, cromoglycates and/or long-acting beta-agonists within 1 week prior to screening and is unable to abstain from them throughout the study.
* Unable to abstain from other medications including non-steroidal anti-inflammatory drugs (NSAIDs), anti-depressant drugs, anti-histamines and anti-asthma (not including steroids), anti-rhinitis or hay fever medication, other than short acting inhaled beta-agonists and paracetamol (up to 4 g per day) for the treatment of minor ailments eg headache from 7 days before screening until the follow-up visit.
* Unable to abstain from medication or supplements that significantly inhibit the cytochrome P450 subfamily enzyme CYP3A4, including ritonavir and ketoconazol from screening and throughout the study.
* Unable to use the DISKHALER and/or DISKUS device correctly.
* History of being unable to tolerate or complete methacholine or allergen challenge tests.
* If, after 2 concurrent administrations of saline during the allergen challenge at screening the subjects still have a fall in FEV1 of greater than 10%.
* Subject is undergoing allergen desensitisation therapy.
* History of sensitivity to any of the study medications (including lactose), or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects who are kept due to regulatory or juridical order in an institution.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-02-16 (Actual); Primary Completion 2009-11-03 (Actual); Study Completion 2009-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Germany (4):
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bareille P, Allen A, Hardes K, Donald A. Effect of repeat inhaled doses of GW870086 on the allergen-induced early and late asthmatic response in subjects with mild asthma. Curr Drug Ther. 2013;8(2)
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 110762 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110762 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110762 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110762 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110762 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110762 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110762 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 24 participants were enrolled from February-2009 to November-2009. ROTADISK™, DISKHALER™ and DISKUS™ were registered trademark product of GlaxoSmithKline.
Pre-assignment Details: Participants with pre-bronchodilator forced expiratory volume in 1 second (FEV1) >65% predicted at Screening, positive wheal and flare reaction (>=3 millimeter) on skin prick testing, early asthmatic response (EAR) and late asthmatic response (LAR) had to include a fall in FEV1 of >=20%, >=15%, respectively from the post saline value were included.
Groups:
- Overall Study: Participants were assigned to take 3 out of the 5 possible treatments for 13 days in a double-blind double dummy design: GW870086 0.25 milligram (mg), 1 mg, 3 mg once daily (OD), active control (fluticasone propionate 0.25 mg bi-daily [BID]) or placebo in accordance with the randomization schedule in each treatment period. All participants received matching placebo during one of the 3 treatment periods. All formulations were prepared in lactose inhalation blend and administered through oral inhalation. GW870086 was provided as ROTADISK, while fluticasone propionate as multi-dose powder inhaler (MDPI). GW870086 was administered via DISKHALER, while fluticasone propionate via DISKUS inhaler. There was a at least 14 days of washout from Day 13 dose.
Period: Overall Study
Arm/Group | Overall Study
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Participants were assigned to take 3 out of the 5 possible treatments for 13 days in a double-blind double dummy design: GW870086 0.25 mg, 1 mg, 3 mg OD, active control (fluticasone propionate 0.25mg BID) or placebo in accordance with the randomization schedule in each treatment period. All participants received matching placebo during one of the 3 treatment periods. All formulations were prepared in lactose inhalation blend and administered through oral inhalation. GW870086 was provided as ROTADISK, while fluticasone propionate as MDPI. GW870086 was administered via DISKHALER, while fluticasone propionate via DISKUS inhaler. There was a at least 14 days of washout from Day 13 dose.
Arm/Group | Overall Study
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.4 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Late Asthmatic Response (LAR): Minimum FEV1 Between 4-10 Hours After Allergen Challenge on Day 13 of Each Treatment Period
Description: Analyzed using a mixed effects model including covariates for participant level Baseline FEV1 and period level Baseline FEV1. Participant level Baseline defined as the mean of Day 1 pre-dose values across periods for each participant and period level Baseline as the difference between the Day 1 pre-dose value and participant level Baseline for each period. Absolute change from saline Baseline was calculated for each participant and time point as value equal to highest challenge value minus highest saline value. Minimum FEV1 over 4-10 hours post allergen challenge was minimum value of all the post-saline time points between 4 to 10 hours (4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5 and 10 hours). The adjusted mean is presented as least square mean (LSM).
Time Frame: 4-10 hours after allergen challenge on Day 13 of each treatment period
Population: The all subject population was used which was defined as all participants who received at least one dose of study medication. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- Placebo: Participants were assigned to take matching placebo of GW870086 or fluticasone propionate for 13 days in accordance with the randomization schedule in each treatment period. All participants received matching placebo during one of the 3 treatment periods. All formulations were prepared in lactose inhalation blend and administered through oral inhalation. Placebo of GW870086 was provided as ROTADISK, while placebo of fluticasone propionate as MDPI. Placebo of GW870086 was administered via DISKHALER, while placebo of fluticasone propionate via DISKUS inhaler. There was a at least 14 days of washout from Day 13 dose.
- GW870086 0.25 mg OD: Participants were assigned to take GW870086 0.25 mg OD for 13 days in accordance with the randomization schedule in each treatment period. All participants received matching placebo during one of the 3 treatment periods. The formulation was prepared in lactose inhalation blend and administered through oral inhalation. GW870086 was provided as ROTADISK and was administered via DISKHALER. There was a at least 14 days of washout from Day 13 dose.
- GW870086 1 mg OD: Participants were assigned to take GW870086 1 mg OD for 13 days in accordance with the randomization schedule in each treatment period. All participants received matching placebo during one of the 3 treatment periods. The formulation was prepared in lactose inhalation blend and administered through oral inhalation. GW870086 was provided as ROTADISK and was administered via DISKHALER. There was at least 14 days of washout from Day 13 dose.
- GW870086 3 mg OD: Participants were assigned to take GW870086 3 mg OD for 13 days in accordance with the randomization schedule in each treatment period. All participants received matching placebo during one of the 3 treatment periods. The formulation was prepared in lactose inhalation blend and administered through oral inhalation. GW870086 was provided as ROTADISK and was administered via DISKHALER. There was at least 14 days of washout from Day 13 dose.
- Fluticasone Propionate 0.25 mg BID: Participants were assigned to take fluticasone propionate 0.25 mg BID for 13 days in accordance with the randomization schedule in each treatment period. All participants received matching placebo during one of the 3 treatment periods. All formulations were prepared in lactose inhalation blend and administered through oral inhalation. Fluticasone propionate was provided as MDPI and administered via DISKUS inhaler. There was at least 14 days of washout from Day 13 dose.
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 22 | 12 | 11 | 12 | 12
Liters | -0.903 [-1.126 to -0.679] | -0.663 [-0.918 to -0.407] | -0.638 [-0.896 to -0.380] | -0.446 [-0.698 to -0.194] | -0.376 [-0.630 to -0.123]
Statistical Analysis 1: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.240, 95% CI 2-sided [0.031 to 0.449], Standard Error of Mean 0.1033
Statistical Analysis 2: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.265, 95% CI 2-sided [0.053 to 0.477], Standard Error of Mean 0.1048
Statistical Analysis 3: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.456, 95% CI 2-sided [0.255 to 0.657], Standard Error of Mean 0.0993
Statistical Analysis 4: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.526, 95% CI 2-sided [0.319 to 0.733], Standard Error of Mean 0.1025

2. Secondary Outcome: LAR: Weighted Mean FEV1 Between 4-10 Hours After Allergen Challenge on Day 13 of Each Treatment Period.
Description: Analyzed using a mixed effects model including covariates for participant level Baseline FEV1 and period level Baseline FEV1. Participant level Baseline was defined as the mean of Day 1 pre-dose values across periods for each participant and period level Baseline as the difference between the Day 1 pre-dose value and participant level Baseline for each period. Absolute change from saline Baseline was calculated for each participant and time point as value equal to highest challenge value minus highest saline value. Weighted mean LAR was calculated for FEV1 over 4-10 hours (4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5 and 10 hours) post allergen challenge using the linear trapezoidal rule. To calculate weighted mean LAR, all FEV1 values recorded after the administration of rescue medication have been set to the last recorded FEV1 value prior to the administration of rescue medication. The adjusted mean is presented as Least square mean (LSM).
Time Frame: 4-10 hours after allergen challenge on Day 13 of each treatment period
Population: All subject population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 22 | 12 | 11 | 12 | 12
Liters | -0.550 [-0.744 to -0.356] | -0.340 [-0.567 to -0.113] | -0.396 [-0.626 to -0.167] | -0.248 [-0.471 to -0.024] | -0.146 [-0.371 to 0.078]
Statistical Analysis 1: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.210, 95% CI 2-sided [0.013 to 0.407], Standard Error of Mean 0.0975
Statistical Analysis 2: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.154, 95% CI 2-sided [-0.046 to 0.354], Standard Error of Mean 0.0988
Statistical Analysis 3: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.303, 95% CI 2-sided [0.113 to 0.492], Standard Error of Mean 0.0937
Statistical Analysis 4: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.404, 95% CI 2-sided [0.209 to 0.599], Standard Error of Mean 0.0966

3. Secondary Outcome: EAR: Minimum FEV1 and Weighted Mean FEV1 Between 0-2 Hours After Allergen Challenge on Day 13 of Each Treatment Period.
Description: Analyzed using a mixed effects model including covariates for participant level Baseline FEV1 and period level Baseline FEV1. Participant level Baseline was defined as the mean of Day 1 pre-dose values across periods for each participant and period level Baseline as the difference between the Day 1 pre-dose value and participant level Baseline for each period. Absolute change from saline Baseline was calculated for each participant and time point as value equal to highest challenge value minus highest saline value. Minimum FEV1 over 0-2 hrs post-allergen challenge (minimum EAR) was the minimum value of all the post-(bolus) allergen challenge. Weighted mean EAR was calculated for FEV1 over 0-2 hours post allergen challenge using the linear trapezoidal rule. It was measured up to and including 2 hours (5, 10, 15, 20, 30, 45 minutes and 1, 1.5 and 2 hours). The adjusted mean is presented as LSM.
Time Frame: 0-2 hours after challenge on Day 13 of each treatment period (approximately 17 weeks)
Population: All subject population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 22 | 12 | 11 | 12 | 12
Liters
  Minimum FEV1 | -1.339 [-1.603 to -1.075] | -1.364 [-1.675 to -1.052] | -1.233 [-1.549 to -0.918] | -1.100 [-1.407 to -0.794] | -0.805 [-1.113 to -0.496]
  Weighted Mean FEV1 | -0.814 [-1.039 to -0.589] | -0.760 [-1.014 to -0.506] | -0.789 [-1.045 to -0.532] | -0.634 [-0.885 to -0.383] | -0.464 [-0.716 to -0.212]
Statistical Analysis 1: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = -0.025, 95% CI 2-sided [-0.302 to 0.253], Standard Error of Mean 0.1372 — Comparison of Minimum FEV1 between Placebo and GW870086 0.25 mg
Statistical Analysis 2: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.106, 95% CI 2-sided [-0.176 to 0.387], Standard Error of Mean 0.1391 — Comparison of Minimum FEV1 between Placebo and GW870086 1 mg
Statistical Analysis 3: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.239, 95% CI 2-sided [-0.028 to 0.506], Standard Error of Mean 0.1319 — Comparison of Minimum FEV1 between Placebo and GW870086 3 mg
Statistical Analysis 4: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.534, 95% CI 2-sided [0.260 to 0.809], Standard Error of Mean 0.1359 — Comparison of Minimum FEV1 between Placebo and fluticasone propionate 0.25 mg BID
Statistical Analysis 5: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.054, 95% CI 2-sided [-0.145 to 0.253], Standard Error of Mean 0.0984 — Comparison of Weighted Mean FEV1 between Placebo and GW870086 0.25 mg
Statistical Analysis 6: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.026, 95% CI 2-sided [-0.176 to 0.228], Standard Error of Mean 0.0998 — Comparison of Weighted Mean FEV1 between Placebo and GW870086 1 mg
Statistical Analysis 7: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.180, 95% CI 2-sided [-0.011 to 0.371], Standard Error of Mean 0.0945 — Comparison of Weighted Mean FEV1 between Placebo and GW870086 3 mg
Statistical Analysis 8: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.350, 95% CI 2-sided [0.153 to 0.548], Standard Error of Mean 0.0978 — Comparison of Weighted Mean FEV1 between Placebo and fluticasone propionate 0.25 mg BID

4. Secondary Outcome: Concentration of Exhaled NO Pre-dose on Day 13 of Each Treatment Period
Description: Exhaled NO concentration data collected on Day 13 (pre-dose) was log transformed and analysed using a mixed effects model including covariates for participant level Baseline FEV1 and period level Baseline FEV1. Participant level Baseline was defined as the mean of Day 1 pre-dose values across periods for each participant and period level Baseline as the difference between the Day 1 pre-dose value and participant level Baseline for each period. The adjusted mean is presented.
Time Frame: Day 13 of each treatment period (approximately 17 weeks)
Population: All subject population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Parts Per Billion
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 24 | 12 | 12 | 11 | 12
Parts Per Billion | 52.91 [46.10 to 60.72] | 37.76 [30.98 to 46.02] | 34.95 [28.97 to 42.16] | 31.18 [25.62 to 37.95] | 23.57 [19.54 to 28.43]
Statistical Analysis 1: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Ratio of adjusted geometric mean = 0.71, 95% CI 2-sided [0.56 to 0.90], Standard Error of Mean 0.116
Statistical Analysis 2: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Ratio of adjusted geometric mean = 0.66, 95% CI 2-sided [0.53 to 0.82], Standard Error of Mean 0.107
Statistical Analysis 3: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Ratio of adjusted geometric mean = 0.59, 95% CI 2-sided [0.47 to 0.74], Standard Error of Mean 0.112
Statistical Analysis 4: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Ratio of adjusted geometric mean = 0.45, 95% CI 2-sided [0.36 to 0.55], Standard Error of Mean 0.107

5. Secondary Outcome: Concentration of Exhaled NO Post-dose on Day 13 of Each Treatment Period
Description: Exhaled NO concentration data collected on Day 13 (2 and 12 hours post-dose) and was measured 3 times at each time point. The outcome was not assessed and data not reported.
Time Frame: Day 13 of each treatment period (approximately 17 weeks)
Population: All subject population. The results were not collected for exhaled NO post-dose on Day 13.
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Adverse Events (AE), Treatment Emergent Adverse Events (TEAE) and Serious Adverse Events (SAE)
Description: An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Time Frame: Up to 17 weeks
Population: All subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 24 | 12 | 12 | 12 | 12
Participants
  TEAE | 4 | 3 | 5 | 1 | 2
  Any AE | 8 | 4 | 7 | 4 | 3
  Any SAE | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Mean Values for Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Participants were required to rest in the supine position for at least 10 minutes before each reading. SBP and DBP was measured on Day 1 (pre-dose and 1 hour post dose), Day 7 (any time post morning dose), Day 13 (pre allergen challenge [pre saline]) and Day 14 (pre and 1 hour post methacholine challenge).
Time Frame: Up to Day 14 of each treatment period (approximately 17 weeks)
Population: All subject population. Only those participants with data available at the indicated time points were analyzed (represented by n=x,x,x,x,x in the category titles).
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 24 | 12 | 12 | 12 | 12
Millimeters of mercury
  DBP-Day 1, Pre dose, n=24,12,12,12,12 | 76.1 (8.63) | 75.8 (9.26) | 74.7 (6.75) | 76.6 (6.58) | 73.7 (6.27)
  DBP-Day 1, 1h Post dose, n=24,12,12,12,12 | 73.8 (7.42) | 72.3 (8.81) | 72.1 (5.84) | 74.5 (4.81) | 73.5 (7.50)
  DBP-Day 7, Post dose, n=23,11,12,12,12 | 74.0 (7.91) | 75.3 (10.30) | 77.3 (5.71) | 74.8 (6.48) | 73.8 (7.31)
  DBP-Day 13, Pre saline, n=24,12,12,12,12 | 76.4 (7.93) | 73.0 (6.97) | 75.0 (7.47) | 74.2 (7.36) | 73.5 (7.74)
  DBP-Day 14, Pre challenge, n=23,12,12,12,12 | 75.6 (8.04) | 74.3 (9.08) | 77.0 (5.01) | 76.0 (8.80) | 74.8 (6.36)
  DBP-Day 14, 1h Post challenge, n=21,11,11,12,12 | 74.3 (5.59) | 72.3 (6.86) | 73.5 (6.53) | 71.3 (7.32) | 72.9 (7.33)
  SBP-Day 1, Pre dose, n=24,12,12,12,12 | 120.8 (12.11) | 119.8 (8.55) | 121.3 (6.53) | 115.8 (8.67) | 117.1 (7.54)
  SBP-Day 1, 1h Post dose, n=24,12,12,12,12 | 123.8 (10.34) | 122.8 (8.14) | 121.5 (6.75) | 118.6 (9.26) | 119.3 (10.75)
  SBP-Day 7, Post dose, n=23,11,12,12,12 | 118.3 (11.53) | 119.3 (7.62) | 119.4 (7.81) | 113.2 (8.77) | 118.7 (5.02)
  SBP-Day 13, Pre saline, n=24,12,12,12,12 | 121.9 (9.21) | 117.6 (7.12) | 118.8 (9.26) | 120.0 (11.80) | 119.2 (11.92)
  SBP-Day 14, Pre challenge, n=23,12,12,12,12 | 119.7 (11.94) | 119.1 (8.43) | 124.5 (10.08) | 116.8 (9.69) | 119.0 (8.61)
  SBP-Day 14, 1h Post challenge, n=21,11,11,12,12 | 123.8 (9.50) | 121.9 (7.23) | 123.7 (7.81) | 117.1 (8.80) | 119.6 (14.22)

8. Secondary Outcome: Mean Values for Heart Rate
Description: Participants were required to rest in the supine position for at least 10 minutes before each reading. Heart rate was measured on Day 1 (pre-dose and 1 hour post dose), Day 7 (any time post morning dose), Day 13 (pre allergen challenge) and Day 14 (pre and 1 hour post methacholine challenge).
Time Frame: Up to Day 14 of each treatment period (approximately 17 weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 24 | 12 | 12 | 12 | 12
Beats per minute
  HR-Day 1, Pre dose, n=24,12,12,12,12 | 64.5 (8.15) | 61.7 (8.50) | 62.8 (8.68) | 60.5 (6.63) | 58.3 (6.37)
  HR-Day 1, 1h Post dose, n=24,12,12,12,12 | 66.3 (8.87) | 68.2 (9.76) | 62.7 (9.33) | 60.1 (6.71) | 62.1 (6.69)
  HR-Day 7, Post dose, n=23,11,12,12,12 | 63.3 (9.52) | 60.9 (9.27) | 64.0 (9.73) | 62.2 (7.88) | 63.7 (8.16)
  HR-Day 13, Pre saline, n=24,12,12,12,12 | 62.5 (7.17) | 62.3 (6.40) | 64.9 (7.96) | 62.3 (8.54) | 64.0 (6.93)
  HR-Day 14, Pre challenge, n=23,12,12,12,12 | 63.7 (7.83) | 64.5 (7.68) | 64.9 (5.12) | 63.1 (9.76) | 62.1 (6.58)
  HR-Day 14, 1h Post challenge, n=21,11,11,12,12 | 67.9 (8.40) | 71.2 (8.30) | 69.7 (8.22) | 66.1 (8.94) | 67.6 (5.60)

9. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Findings
Description: Single 12-lead ECGs were obtained at each time point during the study using an ECG machine that automatically calculated the heart rate and measures PR, QRS, QT, and QTc intervals. It was measured on Day 1 (pre-dose and 1 hour post dose) and Day 14 (pre and 1 hour post methacholine challenge). Participants with normal (Nr), abnormal not clinically significant (ANCS) and abnormal clinically significant (ACS) ECG was presented.
Time Frame: Up to Day 14 of each treatment period (approximately 17 weeks)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 24 | 12 | 12 | 12 | 12
Participants
  D1,Pre dose,Nr,n=24,12,12,12,12 | 20 | 9 | 10 | 11 | 8
  D1,Pre dose,ANCS,n=24,12,12,12,12 | 4 | 3 | 2 | 1 | 4
  D1,Pre dose,ACS,n=24,12,12,12,12 | 0 | 0 | 0 | 0 | 0
  D1,1h Post dose,Nr,n=23,12,12,12,12 | 16 | 7 | 8 | 11 | 9
  D1,1h Post dose,ANCS,n=23,12,12,12,12 | 7 | 5 | 4 | 1 | 3
  D1,1h Post dose,ACS,n=23,12,12,12,12 | 0 | 0 | 0 | 0 | 0
  D14,Pre challenge,Nr,n=24,12,12,12,12 | 19 | 10 | 10 | 12 | 11
  D14,Pre challenge,ANCS,n=24,12,12,12,12 | 5 | 2 | 2 | 0 | 1
  D14,Pre challenge,ACS,n=24,12,12,12,12 | 0 | 0 | 0 | 0 | 0
  D14,1h Post challenge,Nr,n=21,11,11,12,12 | 19 | 10 | 10 | 11 | 11
  D14,1h Post challenge,ANCS,n=21,11,11,12,12 | 2 | 1 | 1 | 1 | 1
  D14,1h Post challenge,ACS,n=21,11,11,12,12 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Change From Baseline in FEV1-allergen Challenge at Each Time Point
Description: A mixed model analysis was performed separately for each planned time point during the allergen challenge on Day 13, from 5 minutes to 10 hour, including covariates for participant level Baseline FEV1 and period level Baseline FEV1. Participant level Baseline was defined as the mean of Day 1 pre-dose values across periods for each participant and period level Baseline as the difference between the Day 1 pre-dose value and participant level Baseline for each period. Absolute change from saline Baseline was calculated for each participant and time point as value equal to highest challenge value minus highest saline value. FEV1 was measured at 5, 10, 15, 20, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5 and 10 hours. The adjusted mean is presented as LSM.
Time Frame: Up to Day 13 of each treatment period (approximately 17 weeks)
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 24 | 12 | 12 | 12 | 12
Liters
  FEV1-5minutes, n=22,12,11,12,12 | -0.785 [-0.945 to -0.626] | -0.765 [-0.971 to -0.558] | -0.713 [-0.933 to -0.493] | -0.565 [-0.766 to -0.363] | -0.437 [-0.639 to -0.234]
  FEV1-10minutes, n=22,12,11,12,12 | -1.077 [-1.320 to -0.834] | -0.913 [-1.202 to -0.625] | -1.026 [-1.318 to -0.734] | -0.833 [-1.116 to -0.549] | -0.583 [-0.869 to -0.298]
  FEV1-15minutes, n=22,12,10,12,12 | -1.182 [-1.444 to -0.919] | -1.157 [-1.478 to -0.837] | -1.039 [-1.377 to -0.702] | -0.927 [-1.240 to -0.614] | -0.682 [-0.997 to -0.367]
  FEV1-20minutes, n=21,12,11,12,12 | -1.238 [-1.486 to -0.991] | -1.170 [-1.473 to -0.867] | -1.144 [-1.451 to -0.837] | -1.005 [-1.301 to -0.709] | -0.666 [-0.965 to -0.367]
  FEV1-30minutes, n=22,12,11,12,12 | -1.201 [-1.480 to -0.921] | -1.212 [-1.533 to -0.891] | -1.143 [-1.467 to -0.819] | -0.982 [-1.298 to -0.666] | -0.713 [-1.031 to -0.395]
  FEV1-45minutes, n=22,12,11,12,12 | -1.048 [-1.331 to -0.765] | -1.031 [-1.361 to -0.701] | -0.983 [-1.317 to -0.649] | -0.754 [-1.079 to -0.429] | -0.667 [-0.994 to -0.340]
  FEV1-1hour, n=22,12,11,12,12 | -0.865 [-1.127 to -0.604] | -0.820 [-1.122 to -0.517] | -0.882 [-1.188 to -0.576] | -0.638 [-0.936 to -0.340] | -0.523 [-0.823 to -0.223]
  FEV1-1.5hours, n=22,12,11,12,12 | -0.541 [-0.778 to -0.304] | -0.496 [-0.767 to -0.225] | -0.523 [-0.797 to -0.249] | -0.337 [-0.604 to -0.069] | -0.323 [-0.592 to -0.054]
  FEV1-2hours, n=22,12,11,12,12 | -0.311 [-0.487 to -0.135] | -0.215 [-0.427 to -0.002] | -0.459 [-0.675 to -0.244] | -0.195 [-0.403 to 0.014] | -0.184 [-0.395 to 0.026]
  FEV1-2.5hours, n=21,12,11,12,12 | -0.165 [-0.306 to -0.024] | -0.120 [-0.290 to 0.051] | -0.251 [-0.424 to -0.077] | -0.138 [-0.306 to 0.029] | -0.107 [-0.275 to 0.061]
  FEV1-3hours, n=22,12,11,12,12 | -0.131 [-0.268 to 0.005] | -0.104 [-0.274 to 0.066] | -0.172 [-0.344 to 0.001] | -0.086 [-0.252 to 0.081] | -0.158 [-0.326 to 0.009]
  FEV1-3.5hours, n=22,12,11,12,12 | -0.184 [-0.330 to -0.039] | -0.143 [-0.324 to 0.038] | -0.164 [-0.348 to 0.020] | -0.111 [-0.288 to 0.067] | -0.093 [-0.272 to 0.086]
  FEV1-4hours, n=22,12,11,12,12 | -0.196 [-0.344 to -0.048] | -0.222 [-0.409 to -0.036] | -0.201 [-0.390 to -0.012] | -0.065 [-0.247 to 0.118] | -0.112 [-0.296 to 0.072]
  FEV1-4.5hours, n=22,12,11,12,12 | -0.341 [-0.515 to -0.166] | -0.201 [-0.418 to 0.015] | -0.228 [-0.448 to -0.008] | -0.137 [-0.349 to 0.076] | -0.091 [-0.305 to 0.123]
  FEV1-5hours, n=22,12,11,12,12 | -0.376 [-0.554 to -0.199] | -0.227 [-0.439 to -0.016] | -0.246 [-0.460 to -0.032] | -0.195 [-0.403 to 0.013] | -0.139 [-0.348 to 0.071]
  FEV1-5.5hours, n=22,12,11,12,12 | -0.394 [-0.583 to -0.206] | -0.310 [-0.534 to -0.086] | -0.401 [-0.628 to -0.174] | -0.216 [-0.437 to 0.004] | -0.079 [-0.301 to 0.143]
  FEV1-6hours, n=22,12,11,12,12 | -0.519 [-0.731 to -0.308] | -0.308 [-0.559 to -0.056] | -0.342 [-0.596 to -0.087] | -0.231 [-0.478 to 0.016] | -0.152 [-0.401 to 0.096]
  FEV1-6.5hours, n=22,12,11,12,12 | -0.528 [-0.721 to -0.335] | -0.366 [-0.598 to -0.135] | -0.393 [-0.627 to -0.158] | -0.245 [-0.472 to -0.018] | -0.167 [-0.396 to 0.062]
  FEV1-7hours, n=22,12,11,12,12 | -0.589 [-0.796 to -0.381] | -0.366 [-0.618 to -0.114] | -0.409 [-0.665 to -0.153] | -0.202 [-0.449 to 0.045] | -0.222 [-0.471 to 0.027]
  FEV1-7.5hours, n=22,12,11,12,12 | -0.587 [-0.803 to -0.372] | -0.403 [-0.674 to -0.132] | -0.442 [-0.717 to -0.166] | -0.216 [-0.481 to 0.050] | -0.163 [-0.430 to 0.104]
  FEV1-8hours, n=22,12,11,12,12 | -0.648 [-0.866 to -0.431] | -0.401 [-0.662 to -0.141] | -0.481 [-0.745 to -0.216] | -0.191 [-0.447 to 0.065] | -0.092 [-0.350 to 0.166]
  FEV1-8.5hours, n=22,12,11,12,12 | -0.668 [-0.892 to -0.443] | -0.423 [-0.699 to -0.148] | -0.446 [-0.725 to -0.167] | -0.158 [-0.428 to 0.112] | -0.075 [-0.347 to 0.197]
  FEV1-9hours, n=22,12,11,12,12 | -0.652 [-0.878 to -0.427] | -0.498 [-0.765 to -0.231] | -0.509 [-0.780 to -0.238] | -0.160 [-0.423 to 0.103] | -0.093 [-0.358 to 0.172]
  FEV1-9.5hours, n=22,12,11,12,12 | -0.660 [-0.891 to -0.430] | -0.485 [-0.750 to -0.221] | -0.473 [-0.740 to -0.205] | -0.246 [-0.507 to 0.015] | -0.139 [-0.401 to 0.124]
  FEV1-10hours, n=22,12,11,12,12 | -0.646 [-0.875 to -0.418] | -0.562 [-0.821 to -0.302] | -0.478 [-0.740 to -0.216] | -0.206 [-0.462 to 0.050] | -0.133 [-0.390 to 0.125]
Statistical Analysis 1: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.021, 95% CI 2-sided [-0.199 to 0.240], Standard Error of Mean 0.1086 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 5 minutes
Statistical Analysis 2: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.164, 95% CI 2-sided [-0.096 to 0.424], Standard Error of Mean 0.1285 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 10 minutes
Statistical Analysis 3: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.024, 95% CI 2-sided [-0.285 to 0.333], Standard Error of Mean 0.1526 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 15 minutes
Statistical Analysis 4: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.069, 95% CI 2-sided [-0.229 to 0.366], Standard Error of Mean 0.1471 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 20 minutes
Statistical Analysis 5: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = -0.011, 95% CI 2-sided [-0.277 to 0.254], Standard Error of Mean 0.1313 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 30 minutes
Statistical Analysis 6: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.016, 95% CI 2-sided [-0.269 to 0.302], Standard Error of Mean 0.1410 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 45 minutes
Statistical Analysis 7: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.046, 95% CI 2-sided [-0.210 to 0.301], Standard Error of Mean 0.1265 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 1 hour
Statistical Analysis 8: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.045, 95% CI 2-sided [-0.178 to 0.268], Standard Error of Mean 0.1102 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 1.5 hours
Statistical Analysis 9: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.096, 95% CI 2-sided [-0.103 to 0.295], Standard Error of Mean 0.0985 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 2 hours
Statistical Analysis 10: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.045, 95% CI 2-sided [-0.121 to 0.212], Standard Error of Mean 0.0826 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 2.5 hours
Statistical Analysis 11: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.027, 95% CI 2-sided [-0.141 to 0.196], Standard Error of Mean 0.0832 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 3 hours
Statistical Analysis 12: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.042, 95% CI 2-sided [-0.138 to 0.221], Standard Error of Mean 0.0888 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 3.5 hours
Statistical Analysis 13: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = -0.027, 95% CI 2-sided [-0.215 to 0.162], Standard Error of Mean 0.0934 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 4 hour
Statistical Analysis 14: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.139, 95% CI 2-sided [-0.076 to 0.354], Standard Error of Mean 0.1065 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 4.5 hours
Statistical Analysis 15: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.149, 95% CI 2-sided [-0.044 to 0.342], Standard Error of Mean 0.0955 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 5 hours
Statistical Analysis 16: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.084, 95% CI 2-sided [-0.119 to 0.288], Standard Error of Mean 0.1005 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 5.5 hours
Statistical Analysis 17: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.212, 95% CI 2-sided [-0.015 to 0.438], Standard Error of Mean 0.1122 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 6 hours
Statistical Analysis 18: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.162, 95% CI 2-sided [-0.051 to 0.374], Standard Error of Mean 0.1051 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 6.5 hours
Statistical Analysis 19: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.222, 95% CI 2-sided [-0.017 to 0.461], Standard Error of Mean 0.1181 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 7 hour
Statistical Analysis 20: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.185, 95% CI 2-sided [-0.089 to 0.458], Standard Error of Mean 0.1355 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 7.5 hours
Statistical Analysis 21: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.247, 95% CI 2-sided [0.007 to 0.487], Standard Error of Mean 0.1187 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 8 hours
Statistical Analysis 22: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.244, 95% CI 2-sided [-0.021 to 0.509], Standard Error of Mean 0.1313 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 8.5 hours
Statistical Analysis 23: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.154, 95% CI 2-sided [-0.086 to 0.394], Standard Error of Mean 0.1189 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 9 hours
Statistical Analysis 24: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.175, 95% CI 2-sided [-0.044 to 0.394], Standard Error of Mean 0.1085 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 9.5 hours
Statistical Analysis 25: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.085, 95% CI 2-sided [-0.122 to 0.292], Standard Error of Mean 0.1024 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at 10 hours
Statistical Analysis 26: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.072, 95% CI 2-sided [-0.155 to 0.300], Standard Error of Mean 0.1125 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 5 minutes
Statistical Analysis 27: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.051, 95% CI 2-sided [-0.213 to 0.314], Standard Error of Mean 0.1303 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 10 minutes
Statistical Analysis 28: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.142, 95% CI 2-sided [-0.176 to 0.461], Standard Error of Mean 0.1572 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 15 minutes
Statistical Analysis 29: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.094, 95% CI 2-sided [-0.208 to 0.396], Standard Error of Mean 0.1494 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 20 minutes
Statistical Analysis 30: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.058, 95% CI 2-sided [-0.212 to 0.327], Standard Error of Mean 0.1332 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 30 minutes
Statistical Analysis 31: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.065, 95% CI 2-sided [-0.224 to 0.354], Standard Error of Mean 0.1430 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 45 minutes
Statistical Analysis 32: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = -0.016, 95% CI 2-sided [-0.276 to 0.243], Standard Error of Mean 0.1283 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 1 hour
Statistical Analysis 33: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.017, 95% CI 2-sided [-0.209 to 0.244], Standard Error of Mean 0.1118 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 1.5 hours
Statistical Analysis 34: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = -0.148, 95% CI 2-sided [-0.350 to 0.053], Standard Error of Mean 0.0998 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 2 hours
Statistical Analysis 35: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = -0.086, 95% CI 2-sided [-0.253 to 0.082], Standard Error of Mean 0.0829 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 2.5 hours
Statistical Analysis 36: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = -0.040, 95% CI 2-sided [-0.211 to 0.130], Standard Error of Mean 0.0843 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 3 hours
Statistical Analysis 37: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.020, 95% CI 2-sided [-0.161 to 0.202], Standard Error of Mean 0.0900 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 3.5 hours
Statistical Analysis 38: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = -0.005, 95% CI 2-sided [-0.196 to 0.186], Standard Error of Mean 0.0947 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 4 hour
Statistical Analysis 39: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.113, 95% CI 2-sided [-0.105 to 0.330], Standard Error of Mean 0.1079 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 4.5 hours
Statistical Analysis 40: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.130, 95% CI 2-sided [-0.065 to 0.326], Standard Error of Mean 0.0968 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 5 hours
Statistical Analysis 41: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = -0.007, 95% CI 2-sided [-0.213 to 0.199], Standard Error of Mean 0.1019 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 5.5 hours
Statistical Analysis 42: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.178, 95% CI 2-sided [-0.052 to 0.407], Standard Error of Mean 0.1138 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 6 hours
Statistical Analysis 43: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.135, 95% CI 2-sided [-0.080 to 0.351], Standard Error of Mean 0.1065 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 6.5 hours
Statistical Analysis 44: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.179, 95% CI 2-sided [-0.062 to 0.421], Standard Error of Mean 0.1198 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 7 hour
Statistical Analysis 45: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.146, 95% CI 2-sided [-0.131 to 0.423], Standard Error of Mean 0.1373 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 7.5 hours
Statistical Analysis 46: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.168, 95% CI 2-sided [-0.075 to 0.411], Standard Error of Mean 0.1203 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 8 hours
Statistical Analysis 47: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.222, 95% CI 2-sided [-0.047 to 0.490], Standard Error of Mean 0.1331 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 8.5 hours
Statistical Analysis 48: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.143, 95% CI 2-sided [-0.100 to 0.387], Standard Error of Mean 0.1206 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 9 hours
Statistical Analysis 49: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.187, 95% CI 2-sided [-0.035 to 0.410], Standard Error of Mean 0.1100 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 9.5 hours
Statistical Analysis 50: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.168, 95% CI 2-sided [-0.042 to 0.378], Standard Error of Mean 0.1039 — Comparison of FEV1 between placebo and GW870086 1 mg OD at 10 hours
Statistical Analysis 51: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.221, 95% CI 2-sided [0.011 to 0.431], Standard Error of Mean 0.1036 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 5 minutes
Statistical Analysis 52: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.244, 95% CI 2-sided [-0.006 to 0.494], Standard Error of Mean 0.1236 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 10 minutes
Statistical Analysis 53: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.255, 95% CI 2-sided [-0.038 to 0.548], Standard Error of Mean 0.1445 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 15 minutes
Statistical Analysis 54: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.233, 95% CI 2-sided [-0.057 to 0.524], Standard Error of Mean 0.1436 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 20 minutes
Statistical Analysis 55: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.219, 95% CI 2-sided [-0.036 to 0.474], Standard Error of Mean 0.1262 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 30 minutes
Statistical Analysis 56: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.294, 95% CI 2-sided [0.019 to 0.568], Standard Error of Mean 0.1355 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 45 minutes
Statistical Analysis 57: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.227, 95% CI 2-sided [-0.019 to 0.473], Standard Error of Mean 0.1216 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 1 hour
Statistical Analysis 58: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.204, 95% CI 2-sided [-0.010 to 0.418], Standard Error of Mean 0.1059 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 1.5 hours
Statistical Analysis 59: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.116, 95% CI 2-sided [-0.075 to 0.308], Standard Error of Mean 0.0947 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 2 hours
Statistical Analysis 60: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.027, 95% CI 2-sided [-0.136 to 0.190], Standard Error of Mean 0.0805 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 2.5 hours
Statistical Analysis 61: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.046, 95% CI 2-sided [-0.116 to 0.208], Standard Error of Mean 0.0801 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 3 hours
Statistical Analysis 62: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.074, 95% CI 2-sided [-0.099 to 0.247], Standard Error of Mean 0.0855 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 3.5 hour
Statistical Analysis 63: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.131, 95% CI 2-sided [-0.051 to 0.313], Standard Error of Mean 0.0900 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 4 hours
Statistical Analysis 64: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.204, 95% CI 2-sided [-0.004 to 0.411], Standard Error of Mean 0.1025 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 4.5 hours
Statistical Analysis 65: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.181, 95% CI 2-sided [-0.004 to 0.367], Standard Error of Mean 0.0918 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 5 hours
Statistical Analysis 66: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.178, 95% CI 2-sided [-0.018 to 0.373], Standard Error of Mean 0.0967 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 5.5 hours
Statistical Analysis 67: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.288, 95% CI 2-sided [0.070 to 0.506], Standard Error of Mean 0.1079 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 6 hours
Statistical Analysis 68: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.283, 95% CI 2-sided [0.079 to 0.488], Standard Error of Mean 0.1011 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 6.5 hours
Statistical Analysis 69: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.386, 95% CI 2-sided [0.157 to 0.616], Standard Error of Mean 0.1137 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 7 hour
Statistical Analysis 70: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.372, 95% CI 2-sided [0.108 to 0.636], Standard Error of Mean 0.1306 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 7.5 hours
Statistical Analysis 71: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.458, 95% CI 2-sided [0.227 to 0.688], Standard Error of Mean 0.1142 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 8 hours
Statistical Analysis 72: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.509, 95% CI 2-sided [0.254 to 0.765], Standard Error of Mean 0.1264 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 8.5 hours
Statistical Analysis 73: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.492, 95% CI 2-sided [0.261 to 0.723], Standard Error of Mean 0.1144 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 9 hours
Statistical Analysis 74: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.414, 95% CI 2-sided [0.203 to 0.625], Standard Error of Mean 0.1042 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 9.5 hours
Statistical Analysis 75: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.440, 95% CI 2-sided [0.241 to 0.639], Standard Error of Mean 0.0984 — Comparison of FEV1 between placebo and GW870086 3 mg OD at 10 hours
Statistical Analysis 76: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.348, 95% CI 2-sided [0.135 to 0.562], Standard Error of Mean 0.1056 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 5 minutes
Statistical Analysis 77: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.494, 95% CI 2-sided [0.237 to 0.751], Standard Error of Mean 0.1273 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 10 minutes
Statistical Analysis 78: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.499, 95% CI 2-sided [0.199 to 0.800], Standard Error of Mean 0.1484 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 15 minutes
Statistical Analysis 79: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.573, 95% CI 2-sided [0.274 to 0.872], Standard Error of Mean 0.1481 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 20 minutes
Statistical Analysis 80: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.488, 95% CI 2-sided [0.225 to 0.751], Standard Error of Mean 0.1303 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 30 minutes
Statistical Analysis 81: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.380, 95% CI 2-sided [0.098 to 0.663], Standard Error of Mean 0.1398 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 45 minutes
Statistical Analysis 82: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.342, 95% CI 2-sided [0.089 to 0.596], Standard Error of Mean 0.1254 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 1 hour
Statistical Analysis 83: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.218, 95% CI 2-sided [-0.003 to 0.439], Standard Error of Mean 0.1094 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 1.5 hours
Statistical Analysis 84: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.127, 95% CI [-0.070 to 0.323], Standard Error of Mean 0.0974 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 2 hours
Statistical Analysis 85: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.058, 95% CI 2-sided [-0.107 to 0.223], Standard Error of Mean 0.0818 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 2.5 hours
Statistical Analysis 86: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = -0.027, 95% CI 2-sided [-0.192 to 0.139], Standard Error of Mean 0.0821 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 3 hours
Statistical Analysis 87: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.091, 95% CI 2-sided [-0.085 to 0.268], Standard Error of Mean 0.0876 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 3.5 hours
Statistical Analysis 88: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.084, 95% CI 2-sided [-0.102 to 0.269], Standard Error of Mean 0.0921 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 4 hour
Statistical Analysis 89: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.249, 95% CI 2-sided [0.038 to 0.461], Standard Error of Mean 0.1050 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 4.5 hours
Statistical Analysis 90: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.238, 95% CI 2-sided [0.047 to 0.429], Standard Error of Mean 0.0945 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 5 hours
Statistical Analysis 91: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.315, 95% CI 2-sided [0.114 to 0.516], Standard Error of Mean 0.0995 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 5.5 hours
Statistical Analysis 92: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.367, 95% CI 2-sided [0.143 to 0.591], Standard Error of Mean 0.1111 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 6 hours
Statistical Analysis 93: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.361, 95% CI 2-sided [0.151 to 0.571], Standard Error of Mean 0.1040 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 6.5 hours
Statistical Analysis 94: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.367, 95% CI 2-sided [0.131 to 0.602], Standard Error of Mean 0.1168 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 7 hour
Statistical Analysis 95: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.424, 95% CI 2-sided [0.155 to 0.694], Standard Error of Mean 0.1336 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 7.5 hours
Statistical Analysis 96: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.556, 95% CI 2-sided [0.319 to 0.793], Standard Error of Mean 0.1174 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 8 hours
Statistical Analysis 97: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.593, 95% CI [0.331 to 0.854], Standard Error of Mean 0.1297 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 8.5 hours
Statistical Analysis 98: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.559, 95% CI 2-sided [0.322 to 0.797], Standard Error of Mean 0.1177 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 9 hours
Statistical Analysis 99: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.522, 95% CI [0.304 to 0.739], Standard Error of Mean 0.1076 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 9.5 hours
Statistical Analysis 100: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.514, 95% CI [0.308 to 0.719], Standard Error of Mean 0.1017 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at 10 hours

11. Secondary Outcome: Mean Laboratory Values for Platelet, White Blood Cells (WBC), Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils
Description: Blood samples for assessment of hematology was collected on Day 1 (pre-dose) and Day 14 (pre methacholine challenge).
Time Frame: Up to Day 14 of each treatment period (approximately 17 weeks)
Population: All subject population. All participants were present at the time of assessment.
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 24 | 12 | 12 | 12 | 12
Giga cells per liter
  Basophils,Day1,pre-dose | 0.027 (0.0123) | 0.025 (0.0117) | 0.022 (0.0094) | 0.016 (0.0090) | 0.021 (0.0079)
  Basophils,Day14,pre-challenge | 0.021 (0.0118) | 0.020 (0.0113) | 0.027 (0.0107) | 0.018 (0.0094) | 0.023 (0.0089)
  Eosinophils,Day1,pre-dose | 0.417 (0.2395) | 0.289 (0.1451) | 0.429 (0.2930) | 0.308 (0.1579) | 0.459 (0.3528)
  Eosinophils,Day14,pre-challenge | 0.516 (0.2579) | 0.411 (0.1399) | 0.482 (0.2291) | 0.320 (0.1587) | 0.346 (0.2143)
  Lymphocytes,Day1,pre-dose | 1.792 (0.5462) | 1.948 (0.4525) | 2.100 (0.6834) | 1.688 (0.4350) | 1.574 (0.3542)
  Lymphocytes,Day14,pre-challenge | 1.676 (0.4461) | 1.872 (0.4693) | 1.771 (0.4827) | 1.599 (0.5361) | 1.619 (0.3474)
  Monocytes,Day1,pre-dose | 0.384 (0.1283) | 0.393 (0.1277) | 0.340 (0.1041) | 0.329 (0.0598) | 0.338 (0.1024)
  Monocytes,Day14,pre-challenge | 0.362 (0.0909) | 0.378 (0.1100) | 0.382 (0.1712) | 0.355 (0.1313) | 0.364 (0.1125)
  Neutrophils,Day1,pre-dose | 3.258 (1.1745) | 3.829 (1.7236) | 2.966 (1.1941) | 2.811 (0.4711) | 3.251 (1.1947)
  Neutrophils,Day14,pre-challenge | 3.572 (1.4247) | 3.209 (0.8137) | 3.557 (1.3102) | 3.182 (0.7059) | 3.288 (1.0353)
  Platelet,Day1,pre-dose | 233.9 (35.20) | 240.3 (42.02) | 247.3 (47.10) | 229.6 (28.27) | 238.8 (51.34)
  Platelet,Day14,pre-challenge | 230.3 (31.03) | 220.3 (28.04) | 230.4 (24.21) | 229.0 (30.64) | 220.8 (33.76)
  WBC,Day1,pre-dose | 5.88 (1.598) | 6.48 (1.582) | 5.86 (1.405) | 5.15 (0.672) | 5.64 (1.439)
  WBC,Day14,pre-challenge | 6.15 (1.865) | 5.89 (1.124) | 6.22 (1.681) | 5.48 (1.008) | 5.64 (1.158)

12. Secondary Outcome: Change From Baseline in FEV1-non Allergen Challenge
Description: Non-allergen challenge FEV1 data was measured on Day 1, 7, 13 and 14. The FEV1 assessments on Day 1 was taken at pre-dose and those on Day 7 was taken post-dose. On Day 13, the pre-allergen challenge FEV1 values was used and on Day 14 the pre-methacholine challenge FEV1 values was used. Absolute change in FEV1 on Day 7, 13 and 14 from pre-dose FEV1 was analyzed separately using a mixed-effects ANOVA model. Period-level Baseline was defined as the difference between the Day 1 pre-dose value and participant-level Baseline for each period, each participant. The change from Baseline was calculated by subtracting the Baseline value from the individual post-randomization value. Post-randomization values refer to assessments performed post dose and after the Baseline assessment. The adjusted mean is presented as LSM.
Time Frame: Up to Day 14 of each treatment period (approximately 17 weeks)
Population: All subject population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 24 | 12 | 12 | 12 | 12
Liters
  FEV1,Day 7,n=23,11,12,12,12 | -0.110 [-0.229 to 0.010] | 0.185 [0.006 to 0.364] | 0.221 [0.054 to 0.387] | 0.187 [0.021 to 0.353] | 0.213 [0.046 to 0.380]
  FEV1,Day 13,n=24,12,12,12,12 | 0.027 [-0.095 to 0.149] | 0.212 [0.046 to 0.378] | 0.108 [-0.055 to 0.270] | 0.283 [0.120 to 0.445] | 0.256 [0.093 to 0.419]
  FEV1,Day 14,n=23,12,12,12,12 | -0.325 [-0.468 to -0.182] | -0.181 [-0.372 to 0.011] | -0.199 [-0.387 to -0.011] | 0.137 [-0.050 to 0.324] | 0.047 [-0.141 to 0.235]
Statistical Analysis 1: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.295, 95% CI [0.086 to 0.503], Standard Error of Mean 0.1038 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at Day 7
Statistical Analysis 2: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.185, 95% CI 2-sided [0.007 to 0.363], Standard Error of Mean 0.0884 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at Day 13
Statistical Analysis 3: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.144, 95% CI 2-sided [-0.062 to 0.351], Standard Error of Mean 0.1026 — Comparison of FEV1 between placebo and GW870086 0.25 mg OD at Day 14
Statistical Analysis 4: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.330, 95% CI 2-sided [0.133 to 0.527], Standard Error of Mean 0.0979 — Comparison of FEV1 between placebo and GW870086 1 mg OD at Day 7
Statistical Analysis 5: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.081, 95% CI 2-sided [-0.092 to 0.253], Standard Error of Mean 0.0856 — Comparison of FEV1 between placebo and GW870086 1 mg OD at Day 13
Statistical Analysis 6: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.126, 95% CI 2-sided [-0.076 to 0.327], Standard Error of Mean 0.1000 — Comparison of FEV1 between placebo and GW870086 1 mg OD at Day 14
Statistical Analysis 7: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.297, 95% CI 2-sided [0.100 to 0.493], Standard Error of Mean 0.0976 — Comparison of FEV1 between placebo and GW870086 3 mg OD at Day 7
Statistical Analysis 8: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.256, 95% CI 2-sided [0.083 to 0.429], Standard Error of Mean 0.0859 — Comparison of FEV1 between placebo and GW870086 3 mg OD at Day 13
Statistical Analysis 9: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Net) = 0.462, 95% CI 2-sided [0.262 to 0.662], Standard Error of Mean 0.0991 — Comparison of FEV1 between placebo and GW870086 3 mg OD at Day 14
Statistical Analysis 10: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.323, 95% CI 2-sided [0.125 to 0.520], Standard Error of Mean 0.0982 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at Day 7
Statistical Analysis 11: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.229, 95% CI 2-sided [0.057 to 0.402], Standard Error of Mean 0.0858 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at Day 13
Statistical Analysis 12: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.372, 95% CI 2-sided [0.172 to 0.572], Standard Error of Mean 0.0991 — Comparison of FEV1 between placebo and fluticasone propionate 0.25 mg BID at Day 14

13. Secondary Outcome: Mean Laboratory Values for Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC)
Description: Blood samples for assessment of hematology was collected on Day 1 (pre-dose) and Day 14 (pre methacholine challenge).
Time Frame: Up to Day 14 of each treatment period (approximately 17 weeks)
Population: All subject population. All participants were present at the time of assessment.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 24 | 12 | 12 | 12 | 12
Grams per liter
  Hemoglobin,Day1,pre-dose | 149.0 (9.04) | 151.8 (7.58) | 147.1 (10.01) | 145.2 (6.52) | 147.2 (6.01)
  Hemoglobin,Day14,pre-challenge | 147.1 (10.16) | 150.3 (10.23) | 148.6 (9.79) | 140.8 (9.11) | 147.4 (8.14)
  MCHC,Day1,pre-dose | 335.0 (5.43) | 335.9 (6.04) | 336.3 (5.74) | 334.6 (7.24) | 336.3 (4.23)
  MCHC,Day14,pre-challenge | 335.7 (4.97) | 335.8 (5.80) | 337.9 (5.73) | 333.5 (5.57) | 335.7 (6.64)

14. Secondary Outcome: Mean Laboratory Values for Hematocrit
Description: Blood samples for assessment of hematology was collected on Day 1 (pre-dose) and Day 14 (pre methacholine challenge).
Time Frame: Up to Day 14 of each treatment period (approximately 17 weeks)
Population: All subject population. All participants were present at the time of assessment.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 24 | 12 | 12 | 12 | 12
Ratio
  Hematocrit,Day1,pre-dose | 0.4445 (0.02631) | 0.4519 (0.02474) | 0.4369 (0.02850) | 0.4341 (0.01919) | 0.4376 (0.02114)
  Hematocrit,Day14,pre-challenge | 0.4383 (0.02929) | 0.4476 (0.03070) | 0.4396 (0.02950) | 0.4225 (0.02418) | 0.4391 (0.02880)

15. Secondary Outcome: Mean Laboratory Values for Mean Corpuscle Hemoglobin (MCH)
Description: Blood samples for assessment of hematology was collected on Day 1 (pre-dose) and Day 14 (pre methacholine challenge).
Time Frame: Up to Day 14 of each treatment period (approximately 17 weeks)
Population: All subject population. All participants were present at the time of assessment.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 24 | 12 | 12 | 12 | 12
Picograms
  MCH,Day1,pre-dose | 30.84 (1.473) | 31.23 (1.577) | 30.93 (1.652) | 30.86 (1.053) | 30.58 (1.652)
  MCH,Day14,pre-challenge | 30.87 (1.512) | 31.19 (1.576) | 30.92 (1.634) | 30.89 (0.961) | 30.57 (1.629)

16. Secondary Outcome: Mean Laboratory Values for Mean Corpuscle Volume (MCV)
Description: Blood samples for assessment of hematology was collected on Day 1 (pre-dose) and Day 14 (pre methacholine challenge).
Time Frame: Up to Day 14 of each treatment period (approximately 17 weeks)
Population: All subject population. All participants were present at the time of assessment.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 24 | 12 | 12 | 12 | 12
Femtoliters
  MCV,Day1,pre-dose | 92.1 (4.87) | 93.0 (4.43) | 92.0 (4.57) | 92.3 (2.96) | 91.0 (5.39)
  MCV,Day14,pre-challenge | 92.0 (4.53) | 93.0 (3.84) | 91.5 (4.42) | 92.8 (2.89) | 91.2 (5.52)

17. Secondary Outcome: Mean Laboratory Values for Reticulocytes
Description: Blood samples for assessment of hematology was collected on Day 1 (pre-dose) and Day 14 (pre methacholine challenge).
Time Frame: Up to Day 14 of each treatment period (approximately 17 weeks)
Population: All subject population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 24 | 12 | 11 | 12 | 12
Trillion cells per liter
  Reticulocytes,Day1,pre-dose | 0.04626 (0.027363) | 0.04708 (0.026433) | 0.04941 (0.027213) | 0.05176 (0.016041) | 0.05268 (0.017560)
  Reticulocytes,Day14,pre-challenge | 0.04574 (0.016707) | 0.05613 (0.026415) | 0.04720 (0.020698) | 0.04565 (0.017335) | 0.05543 (0.029142)

18. Secondary Outcome: Mean Laboratory Values for Albumin and Total Protein
Description: Blood samples for assessment of clinical chemistry was collected on Day 1 (pre-dose) and Day 14 (pre methacholine challenge).
Time Frame: Up to Day 14 of each treatment period (approximately 17 weeks)
Population: All subject population. All participants were present at the time of assessment.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 24 | 12 | 12 | 12 | 12
Grams per liter
  Albumin,Day1,pre-dose | 45.4 (2.41) | 45.5 (2.94) | 45.2 (2.98) | 45.7 (2.23) | 45.3 (3.42)
  Albumin,Day14,pre-challenge | 44.5 (2.47) | 44.5 (2.15) | 44.6 (2.43) | 44.6 (1.73) | 44.8 (2.25)
  Total protein,Day1,pre-dose | 70.6 (3.48) | 71.3 (3.96) | 68.8 (2.80) | 70.0 (3.10) | 70.6 (2.81)
  Total protein,Day14,pre-challenge | 69.3 (3.60) | 69.6 (3.20) | 67.8 (3.01) | 68.2 (3.76) | 69.6 (3.03)

19. Secondary Outcome: Mean Laboratory Values for Alkaline Phosphatase (ALP), Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST) and Gamma Glutamyl Transferase (GGT)
Description: Blood samples for assessment of clinical chemistry was collected on Day 1 (pre-dose) and Day 14 (pre methacholine challenge). Liver safety parameters (ALT and AST) were also assessed on Day 7 (pre-dose).
Time Frame: Up to Day 14 of each treatment period (approximately 17 weeks)
Population: All subject population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: International unit per liter
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 24 | 12 | 12 | 12 | 12
International unit per liter
  ALP,Day1,pre-dose,n=24,12,12,12,12 | 60.8 (15.08) | 61.5 (11.12) | 57.3 (15.03) | 54.6 (18.08) | 64.1 (11.33)
  ALP,Day14,pre-challenge,n=24,12,12,12,12 | 58.8 (14.52) | 61.2 (13.71) | 55.6 (14.64) | 53.3 (17.39) | 63.7 (9.70)
  ALT,Day1,pre-dose,n=24,12,12,12,12 | 20.6 (7.41) | 17.8 (7.72) | 18.9 (5.37) | 17.6 (7.32) | 21.3 (5.90)
  ALT,Day7,pre-dose,n=23,12,12,12,12 | 19.6 (6.28) | 18.8 (7.45) | 19.5 (6.23) | 17.4 (6.88) | 18.7 (4.16)
  ALT,Day14,pre-challenge,n=24,12,12,12,12 | 18.3 (7.83) | 18.2 (7.06) | 18.4 (4.10) | 16.8 (8.16) | 20.3 (5.77)
  AST,Day1,pre-dose,n=24,12,12,12,12 | 21.3 (6.01) | 19.1 (4.50) | 19.4 (3.80) | 19.3 (5.93) | 23.8 (5.42)
  AST,Day7,pre-dose,n=23,12,12,12,12 | 20.1 (4.48) | 19.5 (4.93) | 20.0 (3.69) | 18.7 (4.12) | 20.3 (3.60)
  AST,Day14,pre-challenge,n=24,12,12,12,12 | 18.5 (4.74) | 18.6 (4.72) | 19.3 (3.92) | 17.8 (4.65) | 21.1 (5.16)
  GGT,Day1,pre-dose,n=24,12,12,12,12 | 30.0 (22.30) | 29.4 (14.98) | 25.9 (7.69) | 24.5 (18.25) | 31.5 (19.76)
  GGT,Day14,pre-challenge,n=24,12,12,12,12 | 28.8 (17.64) | 28.3 (13.94) | 24.9 (6.95) | 23.3 (15.77) | 31.1 (19.78)

20. Secondary Outcome: Mean Laboratory Values for Total Bilirubin, Direct Bilirubin and Creatinine
Description: Blood samples for assessment of clinical chemistry was collected on Day 1 (pre-dose) and Day 14 (pre methacholine challenge). Total bilirubin and direct bilirubin were also assessed on Day 7 (pre-dose).
Time Frame: Up to Day 14 of each treatment period (approximately 17 weeks)
Population: All subject population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 24 | 12 | 12 | 12 | 12
Micromoles per liter
  TB,Day1,pre-dose,n=24,12,12,12,12 | 13.7 (7.06) | 13.9 (6.08) | 12.6 (5.50) | 11.8 (2.90) | 14.7 (5.50)
  TB,Day7,pre-dose,n=23,12,12,12,12 | 11.3 (5.18) | 12.5 (6.24) | 11.8 (5.24) | 10.3 (4.29) | 12.6 (5.43)
  TB,Day14,pre-challenge,n=24,12,12,12,12 | 11.4 (3.70) | 11.4 (5.81) | 12.7 (5.99) | 11.5 (4.54) | 11.7 (4.87)
  DB,Day1,pre-dose,n=24,12,12,12,12 | 2.5 (1.44) | 2.5 (1.09) | 2.3 (0.97) | 2.0 (0.74) | 2.5 (1.17)
  DB,Day7,pre-dose,n=23,12,12,12,12 | 2.2 (1.34) | 2.2 (1.47) | 1.9 (0.90) | 1.9 (1.00) | 2.5 (1.09)
  DB,Day14,pre-challenge,n=24,12,12,12,12 | 2.0 (0.86) | 2.0 (1.13) | 1.9 (1.16) | 2.0 (0.85) | 2.3 (0.87)
  Creatinine,Day1,pre-dose,n=24,12,12,12,12 | 90.7 (9.73) | 89.2 (7.91) | 85.8 (10.38) | 89.3 (11.83) | 86.5 (9.89)
  Creatinine,Day14,pre-challenge,n=24,12,12,12,12 | 87.3 (9.46) | 87.2 (13.91) | 84.3 (13.47) | 89.6 (11.91) | 86.8 (10.06)

21. Secondary Outcome: Mean Laboratory Values for Calcium, Glucose, Potassium, Chloride and Sodium
Description: as for outcome 18
Time Frame: Up to Day 14 of each treatment period (approximately 17 weeks)
Population: All subject population. All participants were present at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 24 | 12 | 12 | 12 | 12
Millimoles per liter
  Calcium,Day1,pre-dose | 2.354 (0.0618) | 2.377 (0.0873) | 2.338 (0.0591) | 2.358 (0.0618) | 2.364 (0.0710)
  Calcium,Day14,pre-challenge | 2.355 (0.0896) | 2.343 (0.0568) | 2.327 (0.0627) | 2.324 (0.0562) | 2.334 (0.0566)
  Chloride,Day1,pre-dose | 103.8 (1.84) | 103.7 (2.02) | 103.8 (2.59) | 104.0 (1.21) | 103.8 (2.05)
  Chloride,Day14,pre-challenge | 104.7 (2.42) | 104.5 (1.68) | 104.6 (1.73) | 104.9 (2.39) | 104.4 (1.62)
  Glucose,Day1,pre-dose | 5.10 (0.443) | 5.04 (0.425) | 5.51 (0.950) | 4.87 (0.375) | 5.15 (0.768)
  Glucose,Day14,pre-challenge | 5.18 (0.832) | 5.09 (0.429) | 5.23 (1.052) | 4.98 (0.283) | 5.32 (0.949)
  Potassium,Day1,pre-dose | 4.38 (0.304) | 4.35 (0.224) | 4.28 (0.205) | 4.32 (0.279) | 4.39 (0.250)
  Potassium,Day14,pre-challenge | 4.35 (0.320) | 4.27 (0.257) | 4.20 (0.338) | 4.36 (0.239) | 4.31 (0.375)
  Sodium,Day1,pre-dose | 139.8 (2.04) | 139.2 (2.17) | 139.1 (1.38) | 139.7 (1.83) | 139.4 (1.83)
  Sodium,Day14,pre-challenge | 140.2 (1.93) | 139.3 (2.19) | 140.4 (1.24) | 139.6 (1.51) | 140.3 (2.14)

22. Secondary Outcome: Provocative Concentration of Methacholine Resulting in a 20% Reduction in FEV1 (PC20) on Day 14 of Each Treatment Period.
Description: Methacholine challenge PC20 data the concentration of methacholine to cause >= 20% decrease (that is change <= -20%) in FEV1 compared with saline [Baseline]) was log transformed and analysed using a mixed effects model including covariates for participant level Baseline FEV1 and period level Baseline FEV1. Participant level Baseline was defined as the mean of Day 1 pre-dose values across periods for each participant and period level Baseline as the difference between the Day 1 pre-dose value and participant level Baseline for each period. The PC20 was obtained by linear interpolation (on the log 2 concentration scale) between the lowest concentration of methacholine that caused at least 20% decrease from Baseline and the preceding concentration. The adjusted mean is presented as LSM.
Time Frame: Day 14 of each treatment period (approximately 17 weeks)
Population: All subject population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: milligrams per milliliter
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 19 | 9 | 9 | 11 | 10
milligrams per milliliter | 0.27 [0.18 to 1.53] | 0.22 [0.12 to 1.51] | 0.33 [0.18 to 1.86] | 0.66 [0.38 to 3.20] | 0.95 [0.52 to 5.56]
Statistical Analysis 1: Comparison: Placebo vs GW870086 0.25 mg OD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-1.30 to 0.66], Standard Error of Mean 0.482 — Doubling dose differences, that is a treatment doubling dose difference of 1 indicates that the concentration of methacholine required to cause a 20% fall in FEV1 in one treatment is twice that in the other (log2[2] = 1)
Statistical Analysis 2: Comparison: Placebo vs GW870086 1 mg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.73 to 1.28], Standard Error of Mean 0.495 — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs GW870086 3 mg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 1.28, 95% CI 2-sided [0.36 to 2.19], Standard Error of Mean 0.450 — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Fluticasone Propionate 0.25 mg BID; Test type: Superiority or Other; Mean Difference (Final Values) = 1.79, 95% CI 2-sided [0.84 to 2.75], Standard Error of Mean 0.469 — [estimate comment as in outcome 22, analysis 1]

23. Secondary Outcome: Assessment of Established Markers of Anti-inflammatory Activity in Sputum on Day 14-cell Counts of Eosinophils and Neutrophils
Description: Sputum induction was performed during each treatment period for biomarker analysis 1-2 hour after the methacholine challenge on Day 14. Sputum samples were collected from a minimum of 10 participants in the study.
Time Frame: Day 14 of each treatment period (approximately 17 weeks)
Population: All subject population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 10^4 cells per milliliter of sputum
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 24 | 12 | 12 | 12 | 12
10^4 cells per milliliter of sputum
  Eosinophils,n=17,6,6,4,10 | 0.024 (1175.3) | 0.015 (1038.7) | 0.015 (309.4) | 0.007 (464.2) | 0.008 (222.0)
  Neutrophils,n=17,6,7,4,10 | 0.064 (1115.2) | 0.086 (3070.0) | 0.069 (228.3) | 0.134 (555.9) | 0.053 (280.8)

24. Secondary Outcome: Assessment of Established Markers of Anti-inflammatory Activity in Sputum on Day 14-myeloperoxidase (MPO)
Description: as for outcome 23
Time Frame: Day 14 of each treatment period (approximately 17 weeks)
Population: All subject population. All participants were present at the time of assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 19 | 7 | 8 | 7 | 10
Picograms per milliliter | 260.246 (93.0) | 330.822 (165.6) | 205.906 (73.5) | 287.877 (85.3) | 251.286 (131.0)

25. Secondary Outcome: Assessment of Established Markers of Anti-inflammatory Activity in Sputum on Day 14-interleukin-8 (IL-8)
Description: as for outcome 23
Time Frame: Day 14 of each treatment period (approximately 17 weeks)
Population: All subject population. All participants were present at the time of assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 19 | 7 | 8 | 7 | 10
Nanograms per milliliter | 863.936 (162.7) | 1252.473 (57.9) | 470.412 (64.2) | 408.389 (127.2) | 820.154 (202.6)

26. Secondary Outcome: Assessment of Established Markers of Anti-inflammatory Activity in Sputum on Day 14-total Protein
Description: as for outcome 23
Time Frame: Day 14 of each treatment period (approximately 17 weeks)
Population: All subject population. All participants were present at the time of assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 19 | 7 | 8 | 7 | 10
Micrograms per milliliter | 232.218 (54.8) | 264.893 (40.6) | 193.891 (38.5) | 263.454 (167.9) | 342.683 (122.8)

27. Secondary Outcome: Number of Participants With Established Markers of Anti-inflammatory Activity in Sputum on Day 14-messenger Ribonucleic Acid (mRNA)
Description: Sputum induction was performed during each treatment period for biomarker analysis 1-2 hour after the methacholine challenge on Day 14. Sputum samples were collected from a minimum of 10 participants in the study. The outcome is not assessed.
Time Frame: Day 14 of each treatment period (approximately 17 weeks)
Population: All subject population. A GSK file note, dated 02 April 2009, was used to document that mRNA would no longer be collected from the sputum samples. This was due to the fact that a suitable laboratory could not be identified to carry out the analysis.
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AE and SAE were reported from the start of investigational product and until the follow-up contact (up to 17 weeks)
Description: All subject population used.
Arm/Group | Placebo | GW870086 0.25 mg OD | GW870086 1 mg OD | GW870086 3 mg OD | Fluticasone Propionate 0.25 mg BID
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 8/24 | 4/12 | 7/12 | 4/12 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=24) | GW870086 0.25 mg OD (N=12) | GW870086 1 mg OD (N=12) | GW870086 3 mg OD (N=12) | Fluticasone Propionate 0.25 mg BID (N=12)
Headache (Nervous system disorders) | 3 | 1 | 6 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 3 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.